CLINICAL TRIAL: NCT07366840
Title: A Phase 3, Randomized Advanced Breast Cancer Study Investigating RC48 Combined With Chemotherapy Versus Guideline-recommended Trastuzumab/Inetetamab Plus Chemotherapy in HER2-Positive Patients With Prior TOP1i-ADC Failure
Brief Title: RC48 Combined With Chemotherapy in HER2-Positive Advanced Breast Cancer Patients With Prior TOP1i-ADC Failure
Acronym: BRIGHT
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2510331-7
Record Dates: First submitted 2026-01-14; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HER2-positive Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — disitamab vedotin; Gemcitabine; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disitamab Vedotin plus chemo (Experimental): Participants received Disitamab Vedotin (RC48), 2.0mg/kg intravenously on day 1 of two-week cycle, plus chemotherapy of physician's choice (gemcitabine 1000mg/m2, intravenously on days 1 and 8 of 21-day cycle, or capecitabine, 1000 mg/m2, orally twice daily on days 1-14 of 21-day cycle), with or without guideline-recommended anti-HER2 monoclonal antibody (Trastuzumab or Inetetamab (an analog of trastuzumab), 8 mg/kg loading dose, intravenously, then 6 mg/kg without loading dose, on day 1 of 21-day cycle) until physician's verified progression or unacceptable toxicity.
  Interventions: Drug: Disitamab Vedotin; Drug: Gemcitabine; Drug: Capecitabine; Drug: Inetetamab
- Trastuzumab plus chemo (Experimental): Participants received chemotherapy of physician's choice (gemcitabine 1000mg/m2, intravenously on days 1 and 8 of 21-day cycle, or capecitabine, 1000mg/m2, orally twice daily on days 1-14 of 21-day cycle), with or without guideline-recommended anti-HER2 monoclonal antibody (Trastuzumab or Inetetamab (an analog of trastuzumab), 8 mg/kg loading dose, intravenously, then 6 mg/kg without loading dose, on day 1 of 21-day cycle) until physician's verified progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Capecitabine; Drug: Trastuzumab; Drug: Inetetamab

INTERVENTIONS:
Drug: Disitamab Vedotin — 2.0mg/kg every two weeks
  Other Names: RC48
  Arms: Disitamab Vedotin plus chemo
Drug: Gemcitabine — 1000mg/m2 on days 1 and 8 every three weeks
Drug: Capecitabine — 1000 mg/m2 twice daily on days 1 to14 every three weeks
Drug: Trastuzumab — 6 mg/kg once every three weeks, with an initial loading dose of 8 mg/kg
  Arms: Trastuzumab plus chemo
Drug: Inetetamab — 6 mg/kg once every three weeks, with an initial loading dose of 8 mg/kg

SUMMARY:
The purpose of this study is to assess the safety and efficacy of RC48 (a HER2 antibody drug conjugate with MMAE payload) in combination with gemcitabine or capecitabine (with or without trastuzumab/inetetamab), for treatment of patients with HER2-positive advanced breast cancer (ABC) who have developed disease progression or intolerance to prior therapy with a topoisomerase I inhibitor antibody-drug conjugate (TOP1i-ADC).

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel-controlled, multi-centered, phase 3 clinical study enrolling patients with HER2-positive ABC who have experienced disease progression or intolerance to prior TOP1i-ADC treatment, with ≤ 3 lines of systemic therapy received in the recurrent/metastatic setting. The study consists of two main parts: Part 1: Run-in Phase and Part 2: Randomized Controlled Trial.

Part 1: Run-in Phase The primary objective of the Run-in Phase is to preliminarily verify whether the addition of trastuzumab or inetetamab to the combination regimen of RC48 plus chemotherapy can enhance the anti-tumor efficacy and whether it is associated with any specific toxicities. This phase comprises two regimens, and 30 patients will be randomized 1:1 to receive treatment with either of the two regimens: RC48 plus Gemcitabine or Capecitabine; RC48 plus Gemcitabine or Capecitabine, plus Trastuzumab or Inetetamab.

. Part 2: Randomized Controlled Trial The primary objective of this part is to assess the anti-tumor activity and safety of the optimal regimen identified in Part 1 in patients with HER2-positive ABC who have failed prior TOP1i-ADC treatment. Eligible patients will be stratified and randomized 1:1 to either the experimental group or the control group. 238 patients are expected to be enrolled in Part 2.

Experimental group: RC48 plus Gemcitabine or Capecitabine ± Trastuzumab or Inetetamab.

Control group: Trastuzumab or Inetetamab plus Gemcitabine or Capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged ≥ 18 years.
* Histologically or cytologically confirmed HER2-positive (IHC 3+ or IHC 2+ with positive FISH) advanced breast cancer.
* Disease progression on or intolerance to prior treatment with a topoisomerase I inhibitor-conjugated antibody-drug conjugate (TOP1i-ADC).
* ≤ 3 lines of systemic therapy received in the recurrent or metastatic setting. Prior exposure to only one ADC agent.
* At least one extracranial measurable lesion according to RECIST v1.1 criteria.
* ECOG Performance Status (PS) of 0 or 1.
* Adequate function of major organs, meeting the following criteria:Hematological criteria:Hemoglobin (HB) ≥ 90 g/L (no blood transfusion within 14 days prior);Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L;Platelet count (PLT) ≥ 75 × 10⁹/L.Biochemical criteria:Total Bilirubin (TBIL) ≤ 1.5 × Upper Limit of Normal (ULN); Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3 × ULN; for subjects with liver metastases, ALT and AST ≤ 5 × ULN;Serum Creatinine (Cr) ≤ 1 × ULN, and calculated Creatinine Clearance Rate (Ccr) > 50 mL/min (using the Cockcroft-Gault formula).
* Expected survival ≥ 3 months.
* No prior radiotherapy, chemotherapy, endocrine therapy, molecular targeted therapy or surgery within 3 weeks prior to the start of the study; complete recovery from acute toxicities of previous treatments (if surgery was performed, surgical wounds must be fully healed); no peripheral neuropathy or peripheral neurotoxicity of Grade 1 at most.
* Female subjects with childbearing potential must use a medically approved contraceptive method during the study treatment period and for at least 3 months after the last administration of the study drug.
* Voluntary participation in the study, provision of written informed consent, and good compliance with study procedures and follow-up schedules.

Exclusion Criteria:

* Unstable brain metastases, leptomeningeal metastases, or untreated brain metastases (excluding subjects with treated and stable brain metastases who have been asymptomatic for ≥ 4 weeks).
* A history of arterial or venous thromboembolic events (e.g., cerebrovascular accident including transient ischemic attack, deep vein thrombosis, pulmonary embolism) within 3 years prior to the start of study treatment.
* Uncontrolled systemic diseases, including diabetes mellitus, hypertension, pulmonary fibrosis, acute lung disease, liver cirrhosis, etc.
* Current active infection requiring systemic treatment.
* Failure to recover from toxicities of prior anti-tumor therapy to CTCAE v5.0 Grade 0 or 1 (except for alopecia, hyperpigmentation, or other conditions deemed by the investigator not to increase the risk of study drug administration).
* A history of clinically significant or uncontrolled cardiac diseases, including severe ventricular arrhythmia, congestive heart failure, angina pectoris, or myocardial infarction within 6 months prior.
* Known immediate or delayed hypersensitivity to RC48 or any of its components.
* Pregnant or lactating women.
* A history of other malignancies within 3 years prior (except for bilateral breast cancer with HER2 positivity in both lesions, cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, papillary thyroid carcinoma with favorable prognosis, or carcinoma in situ of the lung or minimally invasive adenocarcinoma with favorable prognosis).
* Any other conditions that, in the investigator's judgment, make the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 268 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2028-01-16 (Estimated); Study Completion 2029-01-16 (Estimated)

PRIMARY OUTCOMES:
Median progression free survival (by investigator) | The observation period for this endpoint is up to 36 months, and will be terminated early upon disease progression or death.
  Progression-Free Survival (PFS), analyzed using the Kaplan-Meier method, is defined as the time from randomization to the first occurrence of disease progression or death, whichever comes first. For subjects without evidence of disease progression or death at the time of analysis, data will be censored at the date of their last tumor assessment.

SECONDARY OUTCOMES:
Objective Response Rate (by investigator) | Baseline at screening and the time of the identification of disease progression, assessed up to 36 months.
  Objective response rate (ORR), defined as best overall response of either complete or partial response based on RECIST 1.1 criteria, will be assessed among participants who have measurable disease at screening and start protocol therapy.
Median overall survival (by investigator) | The observation period for this endpoint will be terminated upon death or if disease progression occurs after 1 year of follow-up.
  Overall Survival (OS), analyzed using the Kaplan-Meier method, is defined as the time from randomization to death from any cause. For participants who remain alive at the time of analysis, data will be censored at the date of last contact or informed consent withdrawal.
Duration of response (by investigator) | The observation period for this endpoint is up to 36 months, and will be terminated early upon disease progression or death.
  Duration of Overall Response (DOR) is defined as the time from the first documentation of meeting the criteria for Complete Response (CR) or Partial Response (PR) to the first date of objectively confirmed disease recurrence, progression, or death from any cause. For disease progression, the reference shall be the smallest tumor measurements recorded since the initiation of treatment.
Disease control rate (by investigator) | The observation period for this endpoint is up to 36 months, and will be terminated early upon disease progression or death.
  Disease control rate (DCR) is defined as the percentage of participants with CR, PR, or stable disease (SD) by investigator per RECIST v1.1.
Adverse events | The observation period for this endpoint is up to 36 months.
  The number of participants who experienced an adverse event (AE) based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms, whether or not considered related to the investigational medicines.